CLINICAL TRIAL: NCT07404189
Title: Evaluation of the Acceptability and Clinical Effectiveness of Augmenting Comprehensive Primary Care-Based Obesity Management With the Nutu™ Digital Health Platform
Brief Title: Augmenting Primary Care-Based Obesity Management With the Nutu™ Digital Health Platform
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Willow Laboratories, Inc. (Unknown)
Responsible Party: Principal Investigator, Drew Sayer, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300015959
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Obesity & Overweight; Cardiovascular Risk Factors
Keywords: intensive behavioral therapy; digital health coaching; weight management
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: Zelen clinical trial design. FLOW patients offered to augment their treatment plan with the Nutu app can accept or decline this addition to their plan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard FLOW Program (Active Comparator): Participants receive the standard 12-month FLOW program including nutrition counseling, physician visits, and behavioral health support.
  Interventions: Behavioral: FLOW Program
- FLOW + Nutu™ Offer (Experimental): Participants receive standard FLOW care and are offered access to the Nutu™ digital health platform, which may be accepted or declined.
  Interventions: Behavioral: FLOW Program; Behavioral: Nutu™ Offer

INTERVENTIONS:
Behavioral: FLOW Program — Participants receive the 12-month FLOW program including nutrition counseling, physician visits, and behavioral health support.
Behavioral: Nutu™ Offer — FLOW patients will receive an offer to add the Nutu™ digital health platform to their FLOW treatment plan, which can be accepted or declined. Nutu™ includes features such as AI-powered digital health coaching and food/exercise tracking.
  Arms: FLOW + Nutu™ Offer

SUMMARY:
This study evaluates the acceptability and clinical effectiveness of integrating the Nutu™ digital health platform into a comprehensive primary care-based behavioral obesity treatment program using a Zelen randomized controlled trial design.

DETAILED DESCRIPTION:
This pragmatic randomized clinical trial is conducted within the established FLOW program, a 12-month multidisciplinary behavioral obesity treatment aligned with USPSTF recommendations. Patients initiating FLOW are randomized to standard care or FLOW augmented with an offer of Nutu™, an AI-powered digital health platform providing behavioral support and self-monitoring tools. Outcomes are collected quarterly over 12 months using routinely collected clinical data.

ELIGIBILITY:
Inclusion Criteria:

* All patients enrolled in the FLOW clinical program are eligible.

Exclusion Criteria:

* Not a patient of the FLOW clinical program at UAB.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Body Weight | Baseline to 12 months
  Difference in body weight change between groups

SECONDARY OUTCOMES:
Nutu™ Acceptance | Baseline
  Percentage of patients who accept Nutu™ when offered
Nutu™ Engagement | Baseline through 12 months
  Number of patient log-ins to the Nutu™ app among those accepting Nutu™

OTHER OUTCOMES:
Waist Circumference | Baseline to 12 months
  Difference in waist circumference change between groups
Body Fat Percentage | Baseline to 12 months
  Difference in body fat percentage change between groups
Blood Pressure | Baseline to 12 months
  Difference in change in blood pressure between groups
LDL Cholesterol | Baseline to 12 months
  Difference in change in LDL Cholesterol between groups
Total Cholesterol | Baseline to 12 months
  Difference in change in total cholesterol between groups
Vertical Jump Height | Baseline to 12 months
  Difference in change in vertical jump height between groups
Grip Strength | Baseline to 12 months
  Difference in change in hand grip strength between groups
Mindfulness | Baseline to 12 months
  Mindfulness Questionnaire. Difference in change in mindfulness between groups.
Resilience | Baseline to 12 months
  Brief Resilience Scale. Difference in change in resilience between groups
Quality of Life | Baseline to 12 months
  Quality of Life Scale. Difference in change in quality of life between groups
Happiness | Baseline to 12 months
  Oxford Happiness Scale. Difference in changes in happiness between groups
Hemoglobin A1c | Baseline to 12 months
  Difference in change in hemoglobin A1c between groups
HDL Cholesterol | Baseline to 12 months
  Difference in change in HDL cholesterol between groups
Triglycerides | Baseline to 12 months
  Difference in change in triglycerides between groups

CONTACTS AND LOCATIONS:
Overall Officials: Drew Sayer, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Hospital - Highlands, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
A fully de-identified dataset will be shared at the time of publication of the primary results of this trial. The dataset will enable other investigators to replicate the primary study analysis.
Supporting Information: SAP, Analytic Code
Time Frame: IDP, SAP, and analytic code will be available upon publication of the primary outcomes manuscript for this trial
Access Criteria: IDP and supporting information will be made available on PubMed Central along with the primary outcomes manuscript.

REFERENCES:
- [Background] Simon GE, Shortreed SM, DeBar LL. Zelen design clinical trials: why, when, and how. Trials. 2021 Aug 17;22(1):541. doi: 10.1186/s13063-021-05517-w. PMID 34404466